CLINICAL TRIAL: NCT02480296
Title: A Phase 1, Double-blind, Randomized, Placebo-controlled, Ascending Multiple Oral Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MYK-461 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Oral Doses of MYK-461 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MyoKardia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MYK461-003
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Healthy
MeSH Terms: interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MYK-461 (Experimental): Oral Tablet x 28 days
  Interventions: Drug: MYK-461
- Placebo (Placebo Comparator): Oral Tablet x 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MYK-461
  Arms: MYK-461
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to establish safety, tolerability, pharmacokinetics and pharmacodynamics of multiple doses of MYK-461 in human subjects. This is a randomized, double-blind, placebo-controlled, sequential group, multiple ascending (oral tablet) dose study in healthy volunteers aged 18-55 years.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index (BMI)
* Normal LVEF
* Normal electrocardiogram (ECG)
* Females must be non pregnant, non lactating and, if sexually active, be using an acceptable birth control method from the time of first dose through 3 months after the last dose of study drug

Exclusion Criteria:

* Any structural abnormalities on echocardiography
* Positive results of HIV test and/or seropositive for HCV or HBV

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the incidence of adverse events | 63 days
  Incidence of adverse events

SECONDARY OUTCOMES:
Determination of pharmacokinetic parameters | 63 days
  maximum concentration (Cmax)
Determination of pharmacokinetic parameters | 63 days
  time of the maximum measured concentration (Tmax)
Determination of pharmacokinetic parameters | 63 days
  area under the concentration time curve (AUC)
Determination of pharmacokinetic parameters | 63 days
  half-life (t1/2)
Characterize pharmacodynamic parameters | 63 days
  echocardiogram assessment
Characterize pharmacodynamic parameters | 63 days
  peak oxygen consumption

CONTACTS AND LOCATIONS:
Overall Officials: Michael Grimm, MD, Study Director — MyoKardia, Inc.
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia